CLINICAL TRIAL: NCT02377609
Title: Cross-validation of the Finger Prick Dried Blood Spot Assay Method With the Established Whole Blood Method for Quantitative Determination of Tacrolimus Blood Concentrations in Transplant Patients
Brief Title: To Validate an Analytical Method to Measure Concentration of Tacrolimus in Blood Taken From Finger Pricks
Status: Terminated | Type: Observational
Why Stopped: DBS method not be validated against the standard of care venepuncture method due to quality of blood sample and variable tacrolimus extraction
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: PMR-EC-1215; 2013-002086-19 (EudraCT Number)
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Validation; Dried Blood Spot; Transplant Patients
Keywords: Dry Blood Spot (DBS); Validation; Tacrolimus; Bioanalytical assay method cross-validation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Dried blood spot and blood collected by venepuncture
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney or Liver Transplant Patients: adult kidney or liver Advagraf® (tacrolimus) recipients
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Advagraf; FK506E

SUMMARY:
The principal aim of this study is to define the relationship between tacrolimus concentrations determined from the finger prick DBS (Dry Blood Spot) method and those determined from blood samples collected by venepuncture in transplant recipients.

DETAILED DESCRIPTION:
This will be a bioanalytical assay method cross-validation study using blood samples donated by up to 100 liver and 100 kidney transplant patients. Subjects who will be attending a routine outpatient follow-up visit will be asked to provide 3 whole blood venepuncture samples (each sample = 3 mL blood) and 3 finger prick DBS blood samples at predose and at 1 and 3 hours postdose. All subjects will be discharged from the study and clinical site at 3 hours postdose. Subjects will derive no benefit from the blood collection procedures and will be paid a predetermined stipend for participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Stable adult transplant recipients aged ≥ 18 years maintained on a once daily Advagraf® based immunosuppressive regimen for the prophylaxis of kidney or liver allograft rejection.

Exclusion Criteria:

* Subjects who are still participating in another clinical study (e.g. attending follow up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable kidney or liver transplant recipient receiving Advagraf® (tacrolimus) therapy
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Cross-validate the dried blood spot (DBS) method by defining the relationship between tacrolimus concentrations determined via DBS method, with those determined using the established and validated whole blood method | 1 day

SECONDARY OUTCOMES:
Compare estimated area under the curve (AUC) values of the DBS and whole blood assay methods using a Bayesian model | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe Ltd.
Locations (6):
- France (4):
  - Site: 7, Clichy
  - Site: 3, Paris
  - Site: 1, Toulouse
  - Site: 5, Villejuif
- United Kingdom (2):
  - Site: 2, Cambridge
  - Site: 6, London